CLINICAL TRIAL: NCT03881657
Title: Sí Texas: Improving Access to Integrated Care for Rio Grande Valley Residents With Severe & Persistent Mental Illness
Brief Title: Reverse Colocated Integrated Care Intervention Among Persons With Severe Persistent Mental Illness at US-Mexico Border
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources in Action, Inc. (Other)
Collaborators: Methodist Healthcare Ministries of South Texas, Inc. (Unknown); Social Innovation Fund (Unknown)
Responsible Party: Principal Investigator, Karen Errichetti, Director, Research and Evaluation, Health Resources in Action, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100001
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Mental Illness Persistent; Chronic Disease; Hypertension; Diabetes; Hypercholesterolemia; Depression; Obesity
Keywords: Integrated Behavioral Health; Reverse Colocation; Integrated Care
MeSH Terms: conditions — Chronic Disease; Hypertension; Diabetes Mellitus; Hypercholesterolemia; Depression; Obesity

STUDY DESIGN:
Intervention Model Description: Treatment group participants were randomized to receive primary care in addition to behavioral health services within a behavioral health setting. Control group participants received behavioral health care services as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group received a reverse colocated integrated behavioral health intervention or usual care
  Interventions: Behavioral: Reverse Colocated Integrated Care
- Control Group (Active Comparator): The control group received behavioral health services only (usual care)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Reverse Colocated Integrated Care — A reverse colocated integrated care model is one where primary care and preventive services are embedded within a behavioral health service setting.
  Arms: Intervention Group
Behavioral: Usual Care — Behavioral health services without primary care or integrated care services
  Arms: Control Group

SUMMARY:
This study evaluated whether patients with severe and persistent mental illness (SPMI) who received coordinated co-located behavioral health and primary care services were more likely to improve health outcomes after 12 months compared to SPMI patients who receive only behavioral health services from the local mental health authority (LMHA) Tropical Texas Behavioral Health (TTBH).The study employed a randomized control trial (RCT) design where intervention participants receiving integrated behavioral health were compared to control participants receiving the usual care provided within an LMHA for SPMI patients. Patients were placed in each group using a randomized number process. Demographic and health outcome data were collected from intervention and control participants at baseline. Health outcome data was subsequently collected at 6-month and 12-month follow-up points.

DETAILED DESCRIPTION:
This study evaluated whether patients with severe and persistent mental illness (SPMI) who received coordinated co-located behavioral health and primary care services were more likely to improve health outcomes after 12 months compared to SPMI patients who receive only behavioral health services from the local mental health authority (LMHA) Tropical Texas Behavioral Health (TTBH).The study employed a randomized control trial (RCT) design where intervention participants receiving integrated behavioral health were compared to control participants receiving the usual care provided within an LMHA for SPMI patients. Patients were placed in each group using a randomized number process. Demographic and health outcome data were collected from intervention and control participants at baseline. Health outcome data was subsequently collected at 6-month and 12-month follow-up points. The primary outcome of interest was systolic blood pressure. Additional secondary outcomes of interest were diastolic blood pressure, HbA1c, BMI, total cholesterol, depressive symptoms, and life functioning. These outcomes were analyzed as continuous variables using linear regression with backward model selection. Longitudinal analyses were also conducted using a likelihood-based approach to general linear mixed models.The intervention and control groups were patients with an SPMI diagnosis over 18 years of age who were not receiving primary care services prior to enrollment and were eligible to receive behavioral health services from TTBH. The participants resided in Cameron or Hidalgo County and had one or more chronic conditions: hypertension (blood pressure of 140/90 mmHg or higher), poorly controlled diabetes (HbA1c over 8.5%), obesity (body mass index of 30.0 or higher), or hypercholesterolemia (total cholesterol level above 200).

ELIGIBILITY:
Inclusion Criteria:

* Reside in Cameron, Hidalgo, or Willacy County
* Have a severe, persistent mental illness as diagnosed by a licensed behavioral health care provider
* Be eligible to receive behavioral health services from TTBH
* Must not be receiving any primary care outside of TTBH (as ascertained via patient self-report)
* Have a diagnosis of one or more chronic conditions:
* Hypertension (blood pressure of 140/90 mmHg or higher)
* Obesity (body mass index of 30.0 or higher)
* Poorly controlled diabetes (HbA1c over 8.5%)
* Hypercholesterolemia (Total cholesterol level above 200)

Exclusion Criteria:

* Not actively suicidal at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Blood pressure | One year
  Blood pressure was measured as a continuous variable (systolic and diastolic) in millimeters of mercury (mmHg).

SECONDARY OUTCOMES:
Blood glucose concentration | One year
  Blood glucose concentration was measured via blood test for HbA1c as a continuous variable
Body mass index | One year
  Height and weight were measured at baseline, and body mass index was calculated
Total cholesterol | One year
  Measured as a continuous variable in milligrams per deciliter
Depressive symptoms | One year
  Measured as a score on the Patient Health Questionnaire-9 tool
Life functioning | One year
  Measured as a score composite of the Adult Needs and Strengths Assessment Tool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Errichetti KS, Flynn A, Gaitan E, Ramirez MM, Baker M, Xuan Z. Randomized Trial of Reverse Colocated Integrated Care on Persons with Severe, Persistent Mental Illness in Southern Texas. J Gen Intern Med. 2020 Jul;35(7):2035-2042. doi: 10.1007/s11606-020-05778-2. Epub 2020 Apr 20. PMID 32314132
- [Derived] Sautter Errichetti K, Ramirez MM, Flynn A, Xuan Z. A reverse colocated integrated care model intervention among persons with severe persistent mental illness at the U.S.-Mexico border: A randomized controlled trial protocol. Contemp Clin Trials Commun. 2019 Nov 12;16:100490. doi: 10.1016/j.conctc.2019.100490. eCollection 2019 Dec. PMID 31872157